CLINICAL TRIAL: NCT00238719
Title: A Double-Blind, Placebo-Controlled, Parallel-Group, Flexible-Dose Study of Venlafaxine ER In Children and Adolescent Outpatients With Social Anxiety Disorder
Brief Title: Study Evaluating Venlafaxine ER in Children and Adolescents With Social Anxiety Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0600B4-389
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2006-05-19 (Estimated); Status verified 2006-05

CONDITIONS: Social Anxiety Disorder
Keywords: Social Anxiety; Children Disorders
MeSH Terms: conditions — Phobia, Social

INTERVENTIONS:
Drug: Venlafaxine ER

SUMMARY:
To determine the anxiolytic efficacy, safety, and tolerability of a flexible-dose of venlafaxine extended release (ER) administered for 16 weeks in the treatment of children and adolescent outpatients with social anxiety disorder (generalized) in a placebo-controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatient
* 8-17 year old
* diagnosis of Social Anxiety Disorder

Exclusion Criteria:

* concomitant psychiatric or medical disorders which interfere with safety or assessment

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 293
Dates: Start 1999-12; Study Completion 2003-06

PRIMARY OUTCOMES:
Final on therapy Social Anxiety Scale-Adolescents and Children (SAS-AC) total score.

SECONDARY OUTCOMES:
Response, defined as a score of 1 (very much improved) or (very improved), on the Clinical Global Impressions-Improvement (CGI-I) scale; Final on therapy Liebowitz Social Anxiety Scale for Children and Adolescents (LSAS-AC) total score.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer